CLINICAL TRIAL: NCT06561126
Title: Engagement of coMmunity Through Participatory Learning and Action for cOntrol and preVEntion of Type II Diabetes and Its Risk Factors [EMPOWER-D]: Cluster Randomized Controlled Trial
Brief Title: Engagement of coMmunity Through Participatory Learning and Action for cOntrol and preVEntion of Type II Diabetes and Its Risk Factors [EMPOWER-D]
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: University of York (Other); Baqai Institute of Diabetology and Endocrinology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMU/DIR/CTU/2024/007; NIHR203248 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2024-08-07; First posted 2024-08-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type II Diabetes Mellitus; Intermediate Hyperglycemia (IHG)
Keywords: Community-Based Participatory; Diabetes Mellitus; Type II Diabetes Mellitus; Intermediate hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The most commonly 2 armed parallel study design would be used to conduct the current study. The 72 cluster will be randomly allocated to one of the two arms. In the rural settings of Pakistan, two districts of the Khyber Pakhtunkhwa province which includes Peshawar and Swabi have been selected. From each cluster, groups will be formed based on the average population size of 1500 per cluster. This ensures the inclusion of diverse settings for a comprehensive study
  The study sites will be selected in a manner that the risk of possible contamination between control and intervention groups is avoided. The intervention group will receive the PLA intervention, while the control arm will only go through assessments i.e., at baseline and end of study.
Masking Description: Non-applicable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participatory, Learning and Action (PLA) Based Intervention (Experimental): Community mobilization will be done via male and female community groups using a PLA Cycle whereby groups themselves identify and priorities problems associated with diabetes and the risk of developing diabetes.Lay facilitators will convene the groups monthly over a period of 18 months, with one meeting per month. A total of 64 groups will be established in each district, each comprising approximately 20-30 participants, covering an eligible population of 250 to 300 individuals. The total number of participants exposed to the intervention, adapted from the DMagic trial in Bangladesh, will be determined based on random selection from the community. The intervention will focus on participatory groups, with separate groups for males and females to ensure inclusivity and encourage participation from high-risk individuals and those with TIIDM.
  Interventions: Behavioral: Participatory, Learning and Action Based Intervention
- Usual Care (No Intervention): The Control Group will not receive the PLA (Participatory Learning and Action) intervention. Study participants in the control group would not be exposed to the training and would be kept in the control group. They would be a group that would receive usual care and routine awareness. However, they will still benefit from the study in several ways. Information about the trial and guidance on who to contact in case of hyperglycemia or intermediate hyperglycemia will be provided. The disease burden in the control area will be monitored, and findings will be included in national and international advocacy and dissemination efforts.

INTERVENTIONS:
Behavioral: Participatory, Learning and Action Based Intervention — The total number of participants exposed to the intervention (adapted from the DMagic trial in Bangladesh) will be determined based on random selection from the community. A PLA-based intervention would be carried out to prepare the Diabetes Mellitus type II patients. The intervention would be carried out for a tentative time of 2 to 3 hours to educate the type II diabetes mellitus. The study participants would be evaluated after 18 months of the intervention. A structured, validated and literature-based assessment checklist will be devised to assess the effectiveness and feasibility of the intervention.
  Arms: Participatory, Learning and Action (PLA) Based Intervention

SUMMARY:
This project aims to adapt, implement, and evaluate Participatory Learning and Action (PLA) based intervention in rural areas of KPK, Pakistan which includes Peshawar and Swabi for TIIDM prevention and control. The pivotal components of this approach include adapting, implementing, and evaluating the PLA-based intervention for the prevention and control of Type II diabetes. These components will be tailored to meet the specific needs of two different settings in Peshawar and Swabi, Pakistan.

Type II Diabetes Mellitus (TIIDM) is considered the fastest-growing health emergency, affecting 537 million adults worldwide. Global projections for the year 2045 suggest that a 12.2% rise in TIIDM is anticipated with an additional 11.4% rise for intermediate hyperglycemia (IHG) [1]. Around 80% of people with TIIDM reside in low-and middle-income countries (LMICs), exhausting the already burdened healthcare system [2]. The intervention "Community groups or mobile phone messaging to prevent and control type 2 diabetes and intermediate hyperglycemia in Bangladesh (DMagic)" has been tested and found effective in the rural context of Bangladesh [1-3]. A full trial will be conducted in the rural areas of Peshawar and Swabi, Pakistan.

It is anticipated that with the use of evidence-based approaches, best practices, and meaningful community participation, PLA is expected to enhance social and behavioural determinants of health and subsequent outcomes. This will further pave the way for the control of other NCDs through a similar focused approach.

DETAILED DESCRIPTION:
The PLA approach has been systematized into a community approach where groups meet together and follow a cycle of activities. This cycle involves problem identification, collaborative strategy planning, implementation, and participatory evaluation. To address community health issues, various strategies including photo voice, group discussions, and role-play have been widely utilized. By leveraging their life experiences, individuals are encouraged to actively participate in these activities, empowering them to identify problems and utilize their skills to develop effective solutions.

Scientific evidence has demonstrated PLA to be a cost-effective technique to increase maternal and neonatal survival in low-resource settings like India and Nepal. Moreover, it increased awareness about birth preparedness, improved newborn care practices, and enhanced male participation in maternal and newborn health.

This study will utilize a community group-based PLA approach to tackle TIIDM (adapted from D-Magic Bangladesh). A cluster randomized controlled trial will be conducted to assess the effectiveness of PLA in addressing TIIDM and pre-diabetes in rural areas of Peshawar and Swabi, Pakistan. The PLA approach is instrumental in improving health outcomes and services by fostering collaborative community efforts and empowering the community. This collaborative approach fosters a sense of unity, inclusivity, and shared responsibility, ultimately contributing to improved health outcomes and the overall well-being of the community. However, despite its significant impact PLA has not been adapted or tested in settings elsewhere for the prevention and control of TIIDM.

Objective:

1. To culturally adapt PLA-based intervention (DMagic) for primary prevention and control of TIIDM in rural communities of Pakistan.
2. To assess the effectiveness of culturally adapted PLA-based intervention (adapted from D-Magic trial Bangladesh) on the two-year cumulative incidence of TIIDM in high-risk individuals and the prevalence of IHG and TIIDM in rural settings.
3. To determine the cost-effectiveness of the adapted DMagic intervention in rural settings of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20 years and above.
* Participants residing in the rural areas of Peshawar and Swabi, Pakistan.
* Individuals willing to participate in the study and provide consent.
* Both individuals with normoglycemia, intermediate hyperglycemia, and diabetes are encouraged to participate.
* Participants who can attend the scheduled meetings and interventions as per the study protocol.

Exclusion Criteria:

* Individuals below the age of 20 years.
* Individuals unwilling to provide consent for participation.
* Participants with severe health conditions that may hinder their active involvement in the study.
* Individuals with a history of non-compliance with medical interventions or research protocols

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12744 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Type 2 Diabetes Mellitus | 18 months
  The study will determine the prevalence of Type 2 Diabetes Mellitus among adults aged 30 years and older by measuring their HbA1c levels at baseline and endline.
Prevalence of Intermediate Hyperglycemia (IHG) | 18 months
  The prevalence of Intermediate Hyperglycemia (IHG) will be assessed using HbA1c and Fasting Blood Glucose (FBG) tests at baseline and endline among adults aged 30 years and older.
2-year cumulative incidence of Type 2 Diabetes Mellitus | 18 months
  The study will calculate the proportion of adults aged 30 years and older with IHG at baseline who progress to Type 2 Diabetes Mellitus within two years.

SECONDARY OUTCOMES:
Blood pressure (BP) | 18 months
  The study will measure and compare mean diastolic and systolic blood pressure at the Baseline and Endline via the Digital BP apparatus.
Prevalence of hypertension | 18 months
  The prevalence of hypertension will be determined based on blood pressure measurements and self-reported antihypertensive medication use among adults aged 30 years and older. Hypertension is defined as BP ≥ 140/90 mmHg or the use of antihypertensive medication.
Abdominal obesity | 18 months
  Use waist-to-hip circumference ratio to assess abdominal obesity separately.
  Waist Circumference: Measured in centimeters.
  Hip Circumference: Measured in centimetres.
  Waist-to-Hip Ratio: Calculated from waist and hip measurements. Abdominal obesity will be assessed by measuring the waist-to-hip circumference ratio among adults aged 20 years and older.
Body mass index (BMI) | 18 months
  The participant's height will be measured in meters while the weight will be measured in kilograms. Weight and height will be combined to report Body mass index (BMI) in kg/m^2. The study will calculate the mean Body mass index BMI among the population.
  The prevalence of weight categories will be determined based on World Health Organization BMI classifications, with severely underweight defined as a BMI less than 16.0 kg/m², underweight as 16.0 to 18.4 kg/m², normal weight as 18.5 to 24.9 kg/m², overweight as 25.0 to 29.9 kg/m², moderately obese as 30.0 to 34.9 kg/m², severely obese as 35.0 to 39.9 kg/m², and morbidly obese as a BMI of 40.0 kg/m² or higher. The results will be reported as the percentage of the population classified into each category.
Prevalence of overweight & obesity | 18 months
  The study will calculate the prevalence of overweight and obesity among the population. Overweight is defined as a Body Mass Index (BMI) of 25.0 to 29.9 kg/m², and obesity is defined as a BMI of 30.0 kg/m² or higher. The results will be reported as the percentage of the population classified into these categories.
Depression | 18 months
  Participants will be screened for depression using the Patient Health Questionnaire-9 at baseline and endline. The Patient Health Questionnaire-9 is a depression screening tool. Higher scores indicate more severe depression. Scores are interpreted as follows:
  0-4: Minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
Body fat composition | 18 months
  Mean body fat percentage will be measured using a Body Fat measuring weighing scale at baseline and endline using a Body Fat (BF) measuring weighing scale
Quality of life of type II diabetes mellitis & Intermediate Hyperglycemia patients | 18 months
  The Quality of Life for type II diabetes mellitus will be measured using the World Health Organization Quality Of Life questionnaire at baseline and endline. World Health Organization Quality Of Life questionaire scores range from 0 to 100, with higher scores indicating a better quality of life.
Anxiety | 18 months
  Participants will be screened for anxiety using the Generalized Anxiety Disorder-7 at baseline and endline. The Generalized Anxiety Disorder-7 is widely recognized and validated for screening and measuring the severity of generalized anxiety disorder. Generalized Anxiety Disorder-7 consists of 7 items, each scored on a scale of 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21. Higher scores indicate more severe anxiety.
  Score Interpretation:
  0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety

OTHER OUTCOMES:
Fruit / vegetable intake | 18 months
  Fruit and vegetable intake frequency was assessed using a Pakistan-validated Food Frequency Questionaire (FFQ) (13) at baseline and endline. The frequency of fruit and vegetable intake will be assessed using a Pakistan-validated Food Frequency Questionnaire (FFQ) and reported as the mean servings per day.
Hemoglobin | 18 months
  Hemoglobin levels were assessed through Complete Blood Count tests at baseline and endline. The hemoglobin levels will be measured in g/dL using a Complete Blood Count test.
Population knowledge about diabetes | 18 months
  Population knowledge about diabetes was assessed using a survey/interview adapted from the DMagic trial at baseline and end-line.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr Zia Ul Haq, MBBS,MPH,PhD, Principal Investigator — Khyber Medical Univeristy Peshawar; Prof. Abdul Basit, MBBS,FRCP, Principal Investigator — Baqai Institute of Diabetology & Endocrinology, Karachi, Pakistan; Zohaib Khan, BDS,MPH,PHD, Principal Investigator — Khyber Medical University; Saima Afaq, MBBS,MPH,PHD, Principal Investigator — University of York
Locations (1):
- Khyber Medical University Peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interested in the stated study area after its proper monitoring. Data or samples shared will be coded, with no PHI included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication.
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators.

REFERENCES:
- [Background] Lam AA, Lepe A, Wild SH, Jackson C. Diabetes comorbidities in low- and middle-income countries: An umbrella review. J Glob Health. 2021 Jul 24;11:04040. doi: 10.7189/jogh.11.04040. eCollection 2021. PMID 34386215
- [Background] Fottrell E, Ahmed N, Morrison J, Kuddus A, Shaha SK, King C, Jennings H, Akter K, Nahar T, Haghparast-Bidgoli H, Khan AKA, Costello A, Azad K. Community groups or mobile phone messaging to prevent and control type 2 diabetes and intermediate hyperglycaemia in Bangladesh (DMagic): a cluster-randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Mar;7(3):200-212. doi: 10.1016/S2213-8587(19)30001-4. Epub 2019 Feb 4. PMID 30733182
- [Background] Lee YL, Lim YMF, Law KB, Sivasampu S. Intra-cluster correlation coefficients in primary care patients with type 2 diabetes and hypertension. Trials. 2020 Jun 16;21(1):530. doi: 10.1186/s13063-020-04349-4. PMID 32546189
- [Background] Martin J, Girling A, Nirantharakumar K, Ryan R, Marshall T, Hemming K. Intra-cluster and inter-period correlation coefficients for cross-sectional cluster randomised controlled trials for type-2 diabetes in UK primary care. Trials. 2016 Aug 15;17:402. doi: 10.1186/s13063-016-1532-9. PMID 27524396
- [Background] Vahedi S. World Health Organization Quality-of-Life Scale (WHOQOL-BREF): Analyses of Their Item Response Theory Properties Based on the Graded Responses Model. Iran J Psychiatry. 2010 Fall;5(4):140-53. PMID 22952508
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Sapra A, Bhandari P, Sharma S, Chanpura T, Lopp L. Using Generalized Anxiety Disorder-2 (GAD-2) and GAD-7 in a Primary Care Setting. Cureus. 2020 May 21;12(5):e8224. doi: 10.7759/cureus.8224. PMID 32582485
- [Background] Ullah I, Islam MS, Ali S, Jamil H, Tahir MJ, Arsh A, Shah J, Islam SMS. Insufficient Physical Activity and Sedentary Behaviors among Medical Students during the COVID-19 Lockdown: Findings from a Cross-Sectional Study in Pakistan. Int J Environ Res Public Health. 2021 Sep 29;18(19):10257. doi: 10.3390/ijerph181910257. PMID 34639559
- [Background] Iqbal R, Haroon MA, Dar FJ, Bilgirami M, Bano G, Khan AH. Validation of a food frequency questionnaire for assessing macronutrient and calcium intake in adult Pakistani population. J Coll Physicians Surg Pak. 2014 Apr;24(4):224-7. PMID 24709231
- [Background] Basit A, Fawwad A, Qureshi H, Shera AS; NDSP Members. Prevalence of diabetes, pre-diabetes and associated risk factors: second National Diabetes Survey of Pakistan (NDSP), 2016-2017. BMJ Open. 2018 Aug 5;8(8):e020961. doi: 10.1136/bmjopen-2017-020961. PMID 30082350
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Derived] Rehman K, Tahir A, Imtiaz S, Khan Z, Afaq S, Khan A, Shah I, Kanaan M, Sanauddin N, Khaleeq N, Abdeali M, Walker S, Ahmed F, Jennings HM, Ali S, Fazid S, Shahab AR, Khattak MI, Zafar R, Basit A, Siddiqi K, Haq ZU. Engagement of coMmunity through Participatory learning and action for cOntrol and preVEntion of type II Diabetes and its Risk factors (EMPOWER-D) - A Protocol for a Cluster Randomised Controlled Trial. BMC Public Health. 2025 Oct 14;25(1):3492. doi: 10.1186/s12889-025-24371-y. PMID 41088044